CLINICAL TRIAL: NCT00662974
Title: A Randomised Double Blind Clinical Trial to Verify if Perineal Massage Increases the Chances of Delivering With an Intact Perineum Comparing the Two Oils. As Secondary Objective, we Will Evaluate the Effects of Perineal Massage on Specific Tear Location, the Severity of Perineal Tears and the Amount of Suture Material Required for Repair
Brief Title: Searching for the Perfect Oil to Protect the Perineum: A Randomized-Controlled, Double-Blind Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Avi Harlev, MD, OBGYN A DEPARTMENT, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: sor468908ctil
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-03

CONDITIONS: Second Stage of Labor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): parturients during the second stage of labor massaged by Wheat Germ Oil
  Interventions: Other: perineal massage with Wheat Germ Oil during the second stage of labor
- B (Experimental): parturients during the second stage of labor massaged by almond oil
  Interventions: Other: perineal massage with almond oil during the second stage of labor

INTERVENTIONS:
Other: perineal massage with Wheat Germ Oil during the second stage of labor — 30 ml of oil applied during labor
  Arms: A
Other: perineal massage with almond oil during the second stage of labor — 30 ml of oil applied during labor
  Arms: B

SUMMARY:
In this study we intend to randomly assign each parturient one of two commonly used oils to be applied during the second stage of labor, one of them containing vitamin E. We will verify if perineal massage increases the chances of delivering with an intact perineum comparing the two oils. As secondary objectives, we will evaluate the effects of perineal massage on specific tear location, the severity of perineal tears and the amount of suture material required for repair.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Term pregnancy

Exclusion Criteria:

* Non-vertex pregnancies
* Multiple pregnancies
* Placenta previa
* Placental abruption
* Intra-uterine infection
* Non progressive labor first stage
* Former operations or surgical procedures in the vagina
* Perineal massage during the weeks before labor

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-12 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
perineal tears vs intact perineum | after delivery

SECONDARY OUTCOMES:
severity of perineal tears amount of suture material required for repair suturing length | after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Delivery Room, Soroka University Medical Center, Beersheba, Israel